CLINICAL TRIAL: NCT03653637
Title: Group (Project Life Force) vs. Individual Suicide Safety Planning RCT
Brief Title: Group ("Project Life Force") vs. Individual Suicide Safety Planning RCT
Acronym: PLF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBB-025-17F; 1I01CX001705-01A1 (NIH)
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Suicide
Keywords: Suicide; Safety Plan; Group Treatment; Veterans
MeSH Terms: conditions — Suicide | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study.
Who Masked: Outcomes Assessor
Masking Description: The individual who evaluates the outcomes of interest will not know the assigned condition of the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Project Life Force (Experimental): A novel, 10-session intervention to enhance currently mandated VA suicide safety planning in a group setting to support its implementation. PLF is a manualized, weekly 90-minute group treatment lasting 10 weeks coinciding with the time frame for enhanced monitoring of Veterans identified as "high-risk". Session content is described in Table 1 (see appendix A). Six of the PLF sessions correspond to a step of the safety plan and teach skills to maximize the use of that particular step of the plan. The use of emotion regulation skills in PLF differs from other DBT interventions in that it focuses primarily on emotion regulation, distraction and developing social support in the specific context of implementing a safety plan. Mindfulness is not covered. PLF is augmented with additional skill modules on physical health management, education pertaining to suicide risk, promoting positive emotion and suicide prevention mobile apps. PLF patients also receive usual care.
  Interventions: Behavioral: Project Life Force
- Treatment-As-Usual (Active Comparator): The comparison condition will be an assessment-only treatment-as-usual (TAU). Research team will track number of individual mental health appointments, SPC outreach contacts, and usage patterns of safety plans. Veterans in both randomized conditions will be receiving the mandated monitoring, outreach, and involvement of SPC staff and clinical team management that constitutes standard VA care for suicidal individuals.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Project Life Force — A novel, 10-session group intervention to enhance currently mandated VA suicide safety planning by involving Veterans who are at high-risk for suicidal. The PLF intervention augments the SSP in a group treatment with skills training, and psychoeducation, to maximize use and effectiveness of the plan. Overall, PLF aims to enhance suicide coping skills, safety planning and connection to others. The primary purpose is to enhance the safety plan with skills training in emotion regulation, building of support and distress tolerance, and enable even acutely-suicidal Veterans to be able to implement the steps of the safety plan.
  Other Names: PLF
  Arms: Project Life Force
Behavioral: Treatment as Usual — The comparison condition will be an assessment-only treatment-as-usual (TAU). Participants in the TAU condition will receive safety planning and specified clinical support, as mandated by their high-risk status.
  Other Names: TAU
  Arms: Treatment-As-Usual

SUMMARY:
The management of suicide risk is a pressing national public health issue especially among Veterans. This grant consists of two arms: the novel treatment and treatment-as-usual. "Project Life Force" (PLF), a novel suicide safety planning group intervention has been developed to provide a mechanism to develop and enhance the Suicide Safety Plan (SSP) over time. PLF, a 10-session, group intervention, combines cognitive behavior therapy (CBT)/dialectical behavior therapy (DBT) skill based, and psychoeducational approaches, to maximize suicide safety planning development and implementation. Veterans revise their plans over several weeks while learning coping, emotion regulation, and interpersonal skills to incorporate into their safety plans.

DETAILED DESCRIPTION:
Worldwide someone dies by suicide every 40 seconds. In the United States, Veterans exhibit significantly higher suicide risk when compared to the general United States population. One in five suicide deaths is a Veteran and in spite of enhanced suicide prevention services in the Veterans Administration (VA), twenty Veterans commit suicide daily. These very concerning numbers demonstrate an urgent need to develop additional, empirically validated interventions for suicidal Veterans.

One component of the VA's coordinated effort to treat high-risk suicidal Veterans, and diminish suicide risk, is through the construction of a Suicide Safety Plan. Considered a best practice, the SSP instructs one to: recognize personal warning signs of suicide; use internal coping strategies; engage social contacts that can offer support and serve as distraction from suicidal thoughts; contact family members or friends who may help resolve a crisis; provide contact information for VA professionals to help and, specify steps for how to make the immediate environment safer. The patient takes the SSP home for his or her use during (or at the onset of) a suicidal crisis. Safety planning is based on the idea that suicide risk fluctuates over time, and aims to prevent suicidal crises from escalating, and stop individuals from acting on their suicidal thoughts and urges. Research suggests creation of the SSP is effective; one study found that Veterans who present to an emergency room show decreased suicide behavior after creating a SSP.

This study aims to fill this treatment gap by examining a novel intervention integrating skills training with safety planning for high risk suicidal Veterans, "Project Life Force" (PLF). The PLF intervention augments the SSP with skills training, and psychoeducation, to maximize use and effectiveness of the plan in a group setting. This intervention's skill instruction is delivered in a group format. Research suggests groups mitigate loneliness and increase a sense of belonging, which is in line with the extensive literature supporting the interpersonal psychological theory (i.e., that those who die by suicide have a low sense of belonging. More recently, reports on the relation of "military unit cohesion" and suicide risk, suggests that increasing unit cohesion may have a protective effect. Overall, PLF aims to enhance suicide coping skills, safety planning and connection to others.

The main objective of this RCT is to examine if Veterans who are at high risk for suicide will benefit from the novel group intervention, PLF, compared to Veterans who receive TAU.The specific aims and hypotheses of PLF are:

Aim 1: To conduct a multi-site randomized clinical trial (RCT) of a group safety planning intervention, "PLF" versus individual safety planning in 265 suicidal Veterans. PLF will be compared with the comparison condition- individual safety planning, the current standard of care, designated as TAU.

Exploratory Aim 2: To test whether increased suicide coping and improved belongingness partially mediates treatment response in PLF>TAU.

Exploratory Aim 3: To test whether group cohesion partially mediates treatment response in PLF.

Exploratory Aim 4: To test whether the change in Safety Plan Quality (post intervention - baseline) is greater PLF>TAU, as well as whether the change in safety plan quality partially mediates treatment response in the follow up period.

Hypothesis A1: Compared to TAU, Veterans who participate in PLF, will demonstrate a decrease in suicidal behavior.

Hypothesis A2: Compared to TAU, Veterans who participate in PLF will show a decrease in depression and hopelessness.

Hypothesis A3: Compared to TAU, Veterans who participate in PLF will have increased compliance and attitudes towards mental health treatment.

ELIGIBILITY:
Inclusion Criteria:

* Discharge from inpatient unit for suicidal ideation or attempts, or placement on the high-risk suicide list maintained by suicide prevention coordinators
* Completion of a safety plan during the past 6 months prior to entry
* Concurrence from the patient's mental health provider for the Veteran to participate in the study and the provider is willing to work with the research team.

Exclusion Criteria:

* Unable to provide informed consent or complete study requirements
* Unable to speak English
* Cognitive difficulties that impair consent capacity
* Unable or unwilling to provide at least one verifiable contact for emergency or tracking purposes
* Unable to attend outpatient group treatment program or tolerate group therapy format
* Active alcohol or opiate dependence requiring medically supervised withdrawal
* Schizophrenia diagnosis
* Participation in another intervention RCT

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne S. Goodman, MD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (2):
- United States (2):
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 294 participants were consented and screened. 87 participants were ineligible and therefore were not randomized, leaving a total of 207 participants randomized to treatment.
Groups:
- Project Life Force: A novel, 10-session intervention to enhance currently mandated VA suicide safety planning in a group setting to support its implementation. PLF is a manualized, weekly 90-minute group treatment lasting 10 weeks coinciding with the time frame for enhanced monitoring of Veterans identified as "high-risk". Six of the PLF sessions correspond to a step of the safety plan and teach skills to maximize the use of that particular step of the plan. The use of emotion regulation skills in PLF differs from other DBT interventions in that it focuses primarily on emotion regulation, distraction and developing social support in the specific context of implementing a safety plan. Mindfulness is not covered. PLF is augmented with additional skill modules on physical health management, education pertaining to suicide risk, promoting positive emotion and suicide prevention mobile apps. PLF patients also receive usual care.
Period: Overall Study
Arm/Group | Project Life Force | Treatment-As-Usual
Started | 101 | 106
Completed | 63 | 68
Not Completed | 38 | 38
Not completed — Death | 1 | 3
Not completed — Lost to Follow-up | 29 | 30
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Project Life Force | Treatment-As-Usual | Total
Number analyzed (Participants) | 101 | 106 | 207
Age, Categorical [Count of Participants; unit: Participants] — Population: The number analyzed differs from the total enrollment of the study because 4 participants did not provide their age and were therefore excluded from the analysis.
  Participants
    number analyzed (Participants) | 99 | 104 | 203
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 90 | 97 | 187
    >=65 years | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The number analyzed differs from the total enrollment of the study because 4 participants did not provide their age and were therefore excluded from this analysis.
  years
    number analyzed (Participants) | 99 | 104 | 203
    (all) | 45.9 (13.8) | 46.4 (14.0) | 46.1 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The number analyzed differs from the total enrollment of the study because 9 participants did not provide their sex and were therefore excluded from the analysis
  Participants
    number analyzed (Participants) | 97 | 101 | 198
    Female | 16 | 12 | 28
    Male | 81 | 89 | 170
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 33 | 69
  Not Hispanic or Latino | 59 | 65 | 124
  Unknown or Not Reported | 6 | 8 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The number analyzed differs from the total enrollment of the study because 6 participants did not provide their sex and were therefore excluded from the analysis.
  Participants
    number analyzed (Participants) | 100 | 102 | 202
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 2 | 2 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 27 | 45 | 72
    White | 45 | 35 | 80
    More than one race | 14 | 12 | 26
    Unknown or Not Reported | 12 | 7 | 19
Region of Enrollment [Number; unit: participants]
  United States | 101 | 106 | 207
Beck Depression Inventory-II [Mean (Standard Deviation); unit: scores on a scale] — The Beck Depression Inventory-II (BDI-II) measures depression symptom severity with 21 items on a Likert scale. It has high internal consistency, construct validity, and test-retest reliability. Each question has a set of at least four possible answer choices ranging in intensity. When the test is scored, a value of 0 to 3 is assigned for each answer, and items are summed for a total score (ranging from 0-63). Higher scores indicate worse depressive severity. Population: Some participants were missing this assessment.
  scores on a scale
    number analyzed (Participants) | 98 | 102 | 200
    (all) | 32.03 (12.45) | 30.90 (15.08) | 31.46 (13.83)
Beck Hopelessness Scale [Mean (Standard Deviation); unit: scores on a scale] — The Beck Hopelessness Scale (BHS) measures hopelessness with 20 binary (true/false) items. Items are recoded so that optimistic beliefs equal 0 and pessimistic beliefs equal 1. Recoded items are summed for a total score (ranging from 0-20), and higher scores indicate more severe hopelessness. The BHS demonstrates excellent internal reliability and external validity. Population: Some participants were missing this assessment.
  scores on a scale
    number analyzed (Participants) | 99 | 102 | 201
    (all) | 10.11 (6.35) | 9.40 (6.61) | 9.75 (6.48)
Suicide-Related Coping Scale [Mean (Standard Deviation); unit: scores on a scale] — The Suicide-Related Coping Scale (SRCS) has 17 items assessing suicide-related coping (knowledge of, and perceived confidence in, using internal coping strategies and external supports to regulate suicidal thoughts and urges). Items are rated on a 5-point scale (Strongly disagree (0) - Strongly agree (4)). All items are summed for a total score (range 0-68), and the first 14 items can also be used for "external coping" and "internal coping" subscales (7 items each; score range 0-28). Higher scores show improved suicide-related coping. The SRCS has acceptable internal and external validity. Population: Some participants were missing this assessment.
  scores on a scale
    number analyzed (Participants) | 99 | 103 | 202
    (all) | 48.30 (10.79) | 49.17 (11.19) | 48.74 (10.98)
Insomnia Severity Index [Mean (Standard Deviation); unit: scores on a scale] — The Insomnia Severity Index (ISI) is a 7-item brief screening measure of insomnia. Items include insomnia severity (falling asleep, staying asleep, and waking too early), satisfaction with sleep, the extent to which sleep difficulties impair daily functioning, how noticeable low quality of life due to sleep difficulties is to others, and distress about sleep difficulties. Item responses range from 0 - 4 and are summed for total scores (range 0-28). Higher scores indicate more severe insomnia. The ISI has good internal consistency and validity for treatment research. Population: Some participants were missing this assessment.
  scores on a scale
    number analyzed (Participants) | 93 | 103 | 196
    (all) | 18.17 (7.26) | 16.98 (7.81) | 17.55 (7.56)
Suicide Intent Scale [Mean (Standard Deviation); unit: scores on a scale] — The Suicide Intent Scale (SIS) measures the retrospective intensity of the wish to die at the time of a suicide attempt with 20 items. Each item is graded in intensity from 0 to 2, and the first 15 items are summed for a total score (ranging from 0 to 30). Higher scores indicate higher suicide intent. The SIS has high inter-rater reliability and internal consistency. Population: The suicide intent scale was only given to participants with specific suicide histories.
  scores on a scale
    number analyzed (Participants) | 84 | 79 | 163
    (all) | 16.74 (4.55) | 16.06 (3.94) | 16.41 (4.27)
Interpersonal Needs Questionnaire-15 [Mean (Standard Deviation); unit: scores on a scale] — The Interpersonal Needs Questionnaire-15 (INQ-15) consists of 15 items assessing thwarted interpersonal needs along two domains: Thwarted Belongingness (TB, nine items) and Perceived Burdensomeness (PB, six items). All items are rated from one (not at all true for me) to seven (very true for me). Six items from the TB subscale are reverse-keyed and reverse-scored. Items are summed for total scores (TB total score range: 9-63 and PB score range: 6-42). Higher scores indicate increased severity of TB and PB. Population: Some participants were missing this assessment.
  scores on a scale
    Thwarted belongingness: number analyzed (Participants) | 96 | 103 | 199
    Thwarted belongingness | 38.64 (11.43) | 39.11 (12.36) | 38.88 (11.89)
    Perceived burdensomeness: number analyzed (Participants) | 96 | 103 | 199
    Perceived burdensomeness | 19.63 (10.73) | 19.57 (11.50) | 19.60 (11.11)
Buss-Perry Aggression Questionnaire [Mean (Standard Deviation); unit: scores on a scale] — The Buss-Perry Aggression Questionnaire (BPAQ) assesses aggression in four domains (anger, hostility, physical aggression, and verbal aggression) with 29 items on a 4-point scale (Extremely uncharacteristic (0) - Extremely characteristic (3)). Items in each domain are summed for domain scores, and higher scores indicate more aggression severity in the respective domain. Total score ranges are: anger: 7-35, hostility: 8-40, physical aggression: 9-45, verbal aggression: 5-25. Population: Some participants were missing this assessment.
  scores on a scale
    Verbal aggression: number analyzed (Participants) | 97 | 103 | 200
    Verbal aggression | 14.64 (4.87) | 15.45 (4.83) | 15.06 (4.85)
    Physical aggression: number analyzed (Participants) | 97 | 103 | 200
    Physical aggression | 25.96 (8.91) | 27.0 (9.02) | 26.50 (8.96)
    Anger: number analyzed (Participants) | 97 | 103 | 200
    Anger | 20.18 (7.23) | 20.27 (6.88) | 20.23 (7.04)
    Hostility: number analyzed (Participants) | 97 | 103 | 200
    Hostility | 25.38 (7.83) | 25.66 (8.22) | 25.53 (8.01)

OUTCOME MEASURES:

1. Primary Outcome: Columbia Suicide Rating Scale (C-SSRS)
Description: Columbia Suicide Rating Scale (C-SSRS) will be used to count prospective or treatment emergent suicidal behaviors. The CSSRS has been used in many treatment trials, and to measure treatment emergent suicidal events during pharmacotherapy.
  C-SSRS contains a subscale on suicidal ideation which is scored from 1-5; higher numbers indicate increased suicidal thinking. The definition of suicide attempt for the primary outcome will consist of any actual suicide attempt, aborted suicide attempt, or interrupted suicide attempt according to the CSSR-S.
Time Frame: Baseline, 3 Month, 6 Month, 12 Month
Population: TAU has 106 participants, but one participant was excluded because we were missing their suicide attempt history information (which the analytic model adjusted for).
Measure: Number; unit: participants with an event
Arm/Group | Project Life Force | Treatment-As-Usual
Number analyzed (Participants) | 101 | 105
participants with an event | 22 | 30
Statistical Analysis 1: Comparison: Project Life Force vs Treatment-As-Usual; Test type: Superiority; p = 0.263, Regression, Cox; This model adjusted for site and lifetime suicide attempt history; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.43 to 1.30] — The HR represents the PLF+TAU group compared to TAU

2. Primary Outcome: Suicidal Behavior by Chart Abstraction
Description: An independent research assessor who is blinded to study condition will complete all outcome assessments. Data for all types of suicidal behavior including suicides, suicide attempts, interrupted attempts, aborted attempts, and preparatory behavior for suicide, will be obtained. The nomenclature and definitions for suicide-related behaviors will follow the Center for Disease Control and Prevention's (CDC) definitions. Suicidal behavior over the 12-month time frame is a cumulative outcome such that detection of suicidal behavior at any of the outcome points, or by any method, leads to a "positive" indication for the suicidal behavior composite.
Time Frame: 12 Month
Population: Data for suicidal behavior measured by the (1) Columbia-Suicide Severity Rating Scale (C-SSRS); Suicidal behavior by Chart Abstraction; and the Death by Suicide by National Death Index Survey Findings were combined into one metric. We mistakenly registered the three outcomes separately, but we intended to use these three data sources to make one suicide attempt variable. As such, we reported all suicidal behavior descriptives and models under the C-SSRS outcome.
Arm/Group | Project Life Force | Treatment-As-Usual
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Death by Suicide by National Death Index Survey Findings
Description: At month 42, each site's research assistant will query the site's state vital statistics registry for all individuals on this list. For all those who are found to be deceased, data will be abstracted pertaining to his/her death and the probability of suicide from the Death Certificate. The 12-month delay in review is necessary because of the well-known lag in recording deaths in state vital statistics registries.
Time Frame: 12 Month
Population: as for outcome 2
Arm/Group | Project Life Force | Treatment-As-Usual
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Beck Depression Inventory-II Change
Description: The Beck Depression Inventory-II (BDI-II) measures depressive severity with 21 items on a Likert scale. It has high internal consistency, construct validity, and test-retest reliability. Each question has a set of at least four possible answer choices ranging in intensity. When the test is scored, a value of 0 to 3 is assigned for each answer, and items are summed for a total score (ranging from 0-63). Higher scores indicate worse depressive severity.
Time Frame: Baseline, 3 Month, 6 Month, 12 Month
Population: Participant drop-out and missing assessment points occurred throughout the duration of the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Project Life Force | Treatment-As-Usual
Number analyzed (Participants) | 98 | 102
score on a scale
  Baseline | 32.03 (12.45) | 30.90 (15.08)
  3 month: number analyzed (Participants) | 61 | 69
  3 month | 23.54 (14.40) | 24.32 (16.04)
  6 month: number analyzed (Participants) | 61 | 63
  6 month | 23.82 (12.52) | 25.19 (17.41)
  12 month: number analyzed (Participants) | 63 | 67
  12 month | 23.87 (12.02) | 21.69 (17.28)
Statistical Analysis 1: Comparison: Project Life Force vs Treatment-As-Usual; Test type: Superiority; p = .72, Mixed Models Analysis — p-value is for the treatment-by-time interaction; The mixed model has a random intercept for participant and is adjusted for site. Time is a linear effect; Slope = -0.07, 95% CI 2-sided [-.43 to .30]; PLF is coded as 1 and TAU is coded as 0

5. Secondary Outcome: Beck Hopelessness Scale Change
Description: The Beck Hopelessness Scale (BHS) measures hopelessness with 20 binary (true/false) items. Items are recoded so that optimistic beliefs equal 0 and pessimistic beliefs equal 1. Recoded items are summed for a total score (ranging from 0-20), and higher scores indicate more severe hopelessness. The BHS demonstrates excellent internal reliability and external validity.
Time Frame: Baseline, 3 Month, 6 Month, 12 Month
Population: Participant drop-out and missing assessment points occurred throughout the duration of the study.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Project Life Force | Treatment-As-Usual
Number analyzed (Participants) | 99 | 102
Score on a scale
  Baseline | 10.11 (6.35) | 9.40 (6.61)
  3-month: number analyzed (Participants) | 62 | 70
  3-month | 7.74 (6.67) | 8.21 (6.59)
  6-month: number analyzed (Participants) | 61 | 63
  6-month | 8.18 (6.38) | 7.67 (7.16)
  12-month: number analyzed (Participants) | 63 | 67
  12-month | 7.48 (6.26) | 7.57 (7.23)
Statistical Analysis 1: Comparison: Project Life Force vs Treatment-As-Usual; Test type: Superiority; p = .23, Mixed Models Analysis — The p-value is for the treatment-by-time interaction; The mixed model has a random intercept for participant and is adjusted for site. Time is a linear effect; Slope = -.10, 95% CI 2-sided [-.43 to .30]; PLF is coded as 1 and TAU is coded as 0

6. Secondary Outcome: Suicide-related Coping Scale Change
Description: The Suicide-Related Coping Scale (SRCS) has 17 items assessing suicide-related coping (knowledge of, and perceived confidence in, using internal coping strategies and external supports to regulate suicidal thoughts and urges). Items are rated on a 5-point scale (Strongly disagree (0) - Strongly agree (4)). All items are summed for a total score (range 0-68), and the first 14 items can also be used for "external coping" and "internal coping" subscales (7 items each; total range 0-28). Higher scores show improved suicide-related coping. The SRCS has acceptable internal and external validity.
Time Frame: Baseline, 3 Month, 6 Month, 12 Month
Population: Participant drop-out and missing assessment points occurred throughout the duration of the study.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Project Life Force | Treatment-As-Usual
Number analyzed (Participants) | 99 | 103
Score on a scale
  Baseline | 48.30 (10.79) | 49.17 (11.19)
  3-month: number analyzed (Participants) | 62 | 70
  3-month | 53.68 (10.67) | 50.09 (14.12)
  6-month: number analyzed (Participants) | 61 | 64
  6-month | 53.15 (10.84) | 49.22 (13.68)
  12-month: number analyzed (Participants) | 63 | 67
  12-month | 53.95 (10.19) | 52.88 (12.15)
Statistical Analysis 1: Comparison: Project Life Force vs Treatment-As-Usual; Test type: Superiority; p = .09, Mixed Models Analysis — The p-value is for the treatment-by-time interaction; The mixed model has a random intercept for participant and is adjusted for site. Time is a linear effect; Slope = .27, 96% CI 2-sided [-.04 to .58]; PLF is coded as 1 and TAU is coded as 0

7. Secondary Outcome: Outpatient Mental Health Treatment Utilization
Description: Outpatient Mental Health Treatment Utilization was quantified using CPRS. The number of outpatient non-PLF mental health visits from the past three months was counted.
Time Frame: 12 Month
Measure: Mean (Standard Deviation); unit: visit count
Arm/Group | Project Life Force | Treatment-As-Usual
Number analyzed (Participants) | 94 | 100
visit count
  Baseline (3-months pre-treatment) | 17.96 (21.50) | 17.53 (15.89)
  6-months post consent | 45.28 (44.40) | 37.82 (30.98)
Statistical Analysis 1: Comparison: Project Life Force vs Treatment-As-Usual; Test type: Superiority; p = .15, Mixed Models Analysis — The p-value is for the treatment-by-time interaction; The mixed model has a random intercept for participant and is adjusted for site; Slope = 1.17, 95% CI 2-sided [-.42 to 2.76] — PLF is coded as 1 and TAU is coded as 0

8. Secondary Outcome: Drug Abuse Screening Test 10 (DAST-10)
Description: The DAST-10 measures drug use over the past twelve months to identify potential drug use disorder with 10 binary items (0/1). Total scores range from 0 to 10. Scores of 0 indicate no problems, 1-2 low-level, 3-5 moderate level, 6-8 substantial level, and 9-10 severe level.
Time Frame: 12 Month
Population: This measure was only administered at the 12-month follow-up. 81 participants filled out the DAST-10 at this assessment point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Project Life Force | Treatment-As-Usual
Number analyzed (Participants) | 35 | 46
Score on a scale | 4.0 (2.83) | 3.57 (3.15)
Statistical Analysis 1: Comparison: Project Life Force vs Treatment-As-Usual; Test type: Superiority; p = .52, t-test, 2 sided; Mean Difference (Final Values) = -.43, 95% CI 2-sided [-1.78 to .91]

9. Secondary Outcome: Alcohol Use Disorders Identification Test-Consumption (AUDIT-C)
Description: The Alcohol Use Disorders Identification Test-Concise (AUDIT-C) is a brief 3-item alcohol screening tool used to identify individuals who may be at risk for hazardous drinking or have an alcohol use disorder. Each item is rated from 0 to 4, and total scores range from 0 - 12. Higher scores indicated an increased likelihood that an individual's drinking is endangering his or her safety.
Time Frame: 12 Month
Population: This measure was only administered at the 12-month follow-up. 124 participants filled out the DAST-10 at this assessment point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Project Life Force | Treatment-As-Usual
Number analyzed (Participants) | 61 | 63
Score on a scale | 1.95 (2.99) | 1.62 (2.56)
Statistical Analysis 1: Comparison: Project Life Force vs Treatment-As-Usual; Test type: Superiority; p = .83, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 188.5 — The estimation parameter statistic provided is the U value from the Mann-Whitney U test

10. Other Pre Specified Outcome: The Group Cohesion Scale-Revised Change
Description: Group cohesion will be measured by the The Group Cohesion Scale-Revised, a 25-item self-report measure that assesses aspects of group cohesion including communication, interaction, member retention, decision making, vulnerability among group members and consistency between group and individual goals with a four-point scale. This scale will be used for participants randomized to the PLF treatment at 3 times points before a group session. The scale demonstrated high validity and reliability in research settings and was found to be sensitive to change in a psychodrama group treatment.
Time Frame: Weeks 1, 5, 10
Population: Data were not collected on this scale when the protocol shifted to virtual treatment due to COVID-19.
Arm/Group | Project Life Force | Treatment-As-Usual
Number analyzed (Participants) | 0 | 0

11. Other Pre Specified Outcome: Interpersonal Needs Questionnaire Change
Description: The Interpersonal Needs Questionnaire-15 (INQ-15) consists of 15 items assessing thwarted interpersonal needs along two domains: Thwarted Belongingness (TB, nine items) and Perceived Burdensomeness (PB, six items). All items are rated from one (not at all true for me) to seven (very true for me). Six items from the TB subscale are reverse-keyed and reverse-scored. Items are summed for total scores (TB total score range: 9-63 and PB score range: 6-42). Higher scores indicate increased severity of TB and PB.
Time Frame: Baseline, 3 Month, 6 Month, 12 Month
Population: Participant drop-out and missing assessment points occurred throughout the duration of the study.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Project Life Force | Treatment-As-Usual
Number analyzed (Participants) | 96 | 103
Score on a scale
  Baseline | 38.64 (11.43) | 39.11 (12.36)
  3-month: number analyzed (Participants) | 60 | 68
  3-month | 33.98 (12.99) | 36.18 (13.85)
  6-month: number analyzed (Participants) | 60 | 61
  6-month | 33.7 (12.79) | 36.20 (13.67)
  12-month: number analyzed (Participants) | 63 | 66
  12-month | 32.29 (12.04) | 34.73 (14.57)
Statistical Analysis 1: Comparison: Project Life Force vs Treatment-As-Usual; Test type: Superiority; p = .24, Mixed Models Analysis — The p-value is for the treatment-by-time interaction; The mixed model has a random intercept for participant and is adjusted for site. Time is a linear effect; Slope = -.22, 95% CI 2-sided [-.58 to .15]; PLF is coded as 1 and TAU is coded as 0

12. Other Pre Specified Outcome: Buss-Perry Aggression Questionnaire Change
Description: The Buss-Perry Aggression Questionnaire (BPAQ) assesses aggression in four domains (anger, hostility, physical aggression, and verbal aggression) with 29 items on a 4-point scale (Extremely uncharacteristic (0) - Extremely characteristic (3)). Items in each domain are summed for domain scores, and higher scores indicate more aggression severity in the respective domain. Total score ranges are: anger: 7-35, hostility: 8-40, physical aggression: 9-45, verbal aggression: 5-25.
Time Frame: Baseline, 3 Month, 6 Month, 12 Month
Population: Participant drop-out and missing assessment points occurred throughout the duration of the study.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Project Life Force | Treatment-As-Usual
Number analyzed (Participants) | 97 | 103
Score on a scale
  Baseline (verbal aggression subscale) | 14.64 (4.87) | 15.45 (4.83)
  3-month (verbal aggression subscale): number analyzed (Participants) | 61 | 70
  3-month (verbal aggression subscale) | 13.56 (4.89) | 15.7 (4.83)
  6-month (verbal aggression subscale): number analyzed (Participants) | 59 | 61
  6-month (verbal aggression subscale) | 13.92 (4.56) | 15.41 (5.17)
  12-month (verbal aggression subscale): number analyzed (Participants) | 63 | 67
  12-month (verbal aggression subscale) | 14.56 (4.74) | 14.36 (4.77)
  Baseline (physical aggression subscale) | 25.96 (8.91) | 27.0 (9.02)
  3-month(physical aggression subscale): number analyzed (Participants) | 61 | 70
  3-month(physical aggression subscale) | 24.61 (8.93) | 27.51 (9.31)
  6-month(physical aggression subscale): number analyzed (Participants) | 59 | 61
  6-month(physical aggression subscale) | 24.15 (7.73) | 26.93 (9.77)
  12-month(physical aggression subscale): number analyzed (Participants) | 63 | 67
  12-month(physical aggression subscale) | 24.35 (9.19) | 25.72 (8.51)
  Baseline (anger subscale) | 20.18 (7.23) | 20.27 (6.88)
  3-month (anger subscale): number analyzed (Participants) | 61 | 70
  3-month (anger subscale) | 19.33 (6.98) | 20.69 (7.32)
  6-month (anger subscale): number analyzed (Participants) | 59 | 61
  6-month (anger subscale) | 19.51 (6.57) | 19.56 (7.49)
  12-month (anger subscale): number analyzed (Participants) | 63 | 67
  12-month (anger subscale) | 18.54 (6.68) | 19.30 (6.59)
  Baseline (hostility subscale) | 25.38 (7.83) | 25.66 (8.22)
  3-month (hostility subscale): number analyzed (Participants) | 61 | 70
  3-month (hostility subscale) | 23.67 (7.69) | 24.33 (8.13)
  6-month (hostility subscale): number analyzed (Participants) | 59 | 61
  6-month (hostility subscale) | 23.86 (6.9) | 23.93 (8.53)
  12-month (hostility subscale): number analyzed (Participants) | 63 | 67
  12-month (hostility subscale) | 23.73 (6.85) | 23.54 (8.71)
Statistical Analysis 1: Comparison: Project Life Force vs Treatment-As-Usual; This analysis concerns the "verbal aggression" subscale; Test type: Superiority; p = .28, Mixed Models Analysis — The p-value is for the treatment-by-time interaction; The mixed model has a random intercept for participant and is adjusted for site. Time is a linear effect; Slope = .07, 95% CI 2-sided [-.06 to .19]; PLF is coded as 1 and TAU is coded as 0
Statistical Analysis 2: Comparison: Project Life Force vs Treatment-As-Usual; This analysis concerns the "physical aggression" subscale; Test type: Superiority; p = .48, Mixed Models Analysis — The p-value is for the treatment-by-time interaction; The mixed model has a random intercept for participant and is adjusted for site. Time is a linear effect; Slope = -.07, 95% CI 2-sided [-.25 to .12] — PLF is coded as 1 and TAU is coded as 0
Statistical Analysis 3: Comparison: Project Life Force vs Treatment-As-Usual; This analysis concerns the "anger" subscale; Test type: Superiority; p = .30, Mixed Models Analysis — The p-value is for the treatment-by-time interaction; The mixed model has a random intercept for participant and is adjusted for site. Time is a linear effect; Slope = -.08, 95% CI 2-sided [-.24 to .07] — PLF is coded as 1 and TAU is coded as 0
Statistical Analysis 4: Comparison: Project Life Force vs Treatment-As-Usual; This analysis concerns the "hostility" subscale; Test type: Superiority; p = .82, Mixed Models Analysis — The p-value is for the treatment-by-time interaction; The mixed model has a random intercept for participant and is adjusted for site. Time is a linear effect; Slope = .02, 95% CI 2-sided [-.17 to .22]; PLF is coded as 1 and TAU is coded as 0

13. Other Pre Specified Outcome: Insomnia Severity Index Change
Description: The Insomnia Severity Index (ISI) is a 7-item brief screening measure of insomnia. Items include insomnia severity (falling asleep, staying asleep, and waking too early), satisfaction with sleep, the extent to which sleep difficulties impair daily functioning, how noticeable low quality of life due to sleep difficulties is to others, and distress about sleep difficulties. Item responses range from 0 - 4 and are summed for total scores (range 0-28). Higher scores indicate more severe insomnia. The ISI has good internal consistency and validity for treatment research.
Time Frame: Baseline, 3 Month, 6 Month, 12 Month
Population: Participant drop-out and missing assessment points occurred throughout the duration of the study.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Project Life Force | Treatment-As-Usual
Number analyzed (Participants) | 93 | 103
Score on a scale
  Baseline | 18.17 (7.26) | 16.98 (7.81)
  3-month: number analyzed (Participants) | 58 | 68
  3-month | 14.59 (8.46) | 14.88 (8.15)
  6-month: number analyzed (Participants) | 60 | 62
  6-month | 13.63 (8.08) | 15.15 (8.36)
  12-month: number analyzed (Participants) | 63 | 64
  12-month | 13.94 (6.60) | 13.63 (8.81)
Statistical Analysis 1: Comparison: Project Life Force vs Treatment-As-Usual; Test type: Superiority; p = .41, Mixed Models Analysis — The p-value is for the treatment-by-time interaction; The mixed model has a random intercept for participant and is adjusted for site. Time is a linear effect; Slope = -.08, 95% CI 2-sided [-.27 to .11] — PLF is coded as 1 and TAU is coded as 0

14. Other Pre Specified Outcome: Beck Lethality Scale Change
Description: The Beck Lethality Scale (BLS) is an interview-administered measure of medical lethality of a suicide attempt for eight possible methods (i.e., coma-producing drugs, non-coma-producing drugs, shooting, burning, drowning, cutting, jumping, and hanging). The BLS was used following suicidal behavior over the full study duration. Each item (i.e., each method) is rated from "0" (none or minimal damage) to "10" (death) based on an examination of the patient's physical condition on admission, review of the medical charts, and consultation with the attending physician. Higher scores on each method indicate higher lethality for that method. The highest lethality rating across all of the eight methods (none or minimal damage to death) was used as a total score.
Time Frame: 12 Month
Population: Number of people who had a suicide attempt (actual attempt) over the study course, excluding baseline attempts, and filled out the Beck Lethality Scale about these attempts.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Project Life Force | Treatment-As-Usual
Number analyzed (Participants) | 8 | 18
score on a scale | 4.41 (4.10) | 3.36 (4.45)
Statistical Analysis 1: Comparison: Project Life Force vs Treatment-As-Usual; Test type: Superiority; p = .67, Mixed Models Analysis — The p-value is for the treatment-by-time interaction; The mixed model has a random intercept for participant and is adjusted for site. Time is a linear effect; Slope = -.13, 95% CI 2-sided [-.68 to .48] — PLF is coded as 1 and TAU is coded as 0

15. Other Pre Specified Outcome: Beck Suicide Intent Scale Change
Description: The Suicide Intent Scale (SIS) measures the retrospective intensity of the wish to die at the time of a suicide attempt with 20 items. Each item is graded in intensity from 0 to 2, and the first 15 items are summed for a total score (ranging from 0 to 30). Higher scores indicate higher suicide intent. The SIS has high inter-rater reliability and internal consistency.
Time Frame: Baseline, 3 Month, 6 Month, 12 Month
Population: Participant drop-out and missing assessment points occurred throughout the duration of the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Project Life Force | Treatment-As-Usual
Number analyzed (Participants) | 101 | 106
score on a scale
  Baseline: number analyzed (Participants) | 84 | 79
  Baseline | 16.74 (4.55) | 16.06 (3.94)
  3-month: number analyzed (Participants) | 7 | 12
  3-month | 16.71 (4.42) | 16.00 (3.57)
  6-month: number analyzed (Participants) | 4 | 7
  6-month | 15.25 (7.27) | 15.14 (4.67)
  12-month: number analyzed (Participants) | 7 | 10
  12-month | 3.23 (2.41) | 17.30 (16.14)

16. Other Pre Specified Outcome: Ohio State University Traumatic Brain Injury Identification Method
Description: The Ohio State University Traumatic Brain Injury Identification Method is a standardized, 3-5-minute structured interview designed elicit a person's lifetime history of TBI.
Time Frame: Baseline
Population: This measure was used for the study's eligibility criteria and was not intended to be an outcome measure.
Arm/Group | Project Life Force | Treatment-As-Usual
Number analyzed (Participants) | 0 | 0

17. Other Pre Specified Outcome: Mini International Neuropsychiatric Interview
Description: The Mini International Neuropsychiatric Interview (MINI) is a structured diagnostic interview that assesses the presence of psychiatric disorders according to DSM-IV or ICD-10 criteria, with good interrater and test-retest reliability. The MINI was used to determine psychiatric diagnoses (lifetime and current).
Time Frame: Baseline
Population: This measure was used for the study's eligibility criteria and was not intended to be an outcome measure.
Arm/Group | Project Life Force | Treatment-As-Usual
Number analyzed (Participants) | 0 | 0

18. Other Pre Specified Outcome: Mini Mental State Exam
Description: The Mini Mental State Exam is a questionnaire used to measure cognitive impairment. This scale has good validity and construct validity and will be used to examine if participants are cognitively able to participate in the study.
Time Frame: Baseline
Population: This measure was used for the study's eligibility criteria and was not intended to be an outcome measure.
Arm/Group | Project Life Force | Treatment-As-Usual
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from participant consent date through study completion, average of one year.
Groups:
- Project Life Force: A novel, 10-session intervention to enhance VA suicide safety planning in a group setting. PLF is a manualized, weekly 90-minute treatment lasting 10 weeks coinciding with the time frame for enhanced monitoring of Veterans identified as "high-risk". Session content is described in Table 1 (see appendix A). Six PLF sessions correspond to steps of the safety plan and teach skills maximizing use of each step of the plan. Emotion regulation skills in PLF differ from other DBT interventions in focusing primarily on emotion regulation, distraction and developing social support in the specific context of implementing a safety plan. Mindfulness is not covered. PLF is augmented with additional skill modules on physical health management, education pertaining to suicide risk, promoting positive emotion and suicide prevention mobile apps. PLF patients also receive usual care. A novel,10-session group intervention enhancing currently mandated VA suicide safety planning by involving Veterans who are at high-risk for suicide. PLF intervention augments the SSP in a group treatment with skills training, and psychoeducation, to maximize use and effectiveness of the plan. Overall, PLF aims to enhance suicide coping skills, safety planning and connection to others. The primary purpose is to enhance the safety plan with skills training in emotion regulation, building of support and distress tolerance, and enable even acutely-suicidal Veterans to be able to implement the steps of the safety plan.
Arm/Group | Project Life Force | Treatment-As-Usual
All-Cause Mortality (participants affected / at risk) | 1/101 | 3/106
Serious Adverse Events (participants affected / at risk) | 31/101 | 29/106
Other Adverse Events (participants affected / at risk) | 8/101 | 4/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Project Life Force (N=101) | Treatment-As-Usual (N=106)
Hospitalized inpatient psych unit (Psychiatric disorders) | 23 (23) | 20 (20)
Inpatient Psychiatric Hospitalization (Psychiatric disorders) | 21 (27) | 19 (21)
Suicide attempt without medical intervention (Psychiatric disorders) | 3 (4) | 3 (4)
Heart Failure (Cardiac disorders) | 1 (4) | 0 (0)
Emergency Department visit for rib pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Emergency Department visit for orthopedic concerns (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Medical hospitalization (unspecified) (General disorders) | 0 (0) | 1 (1)
Hospitalized following motor vehicle accident (General disorders) | 0 (0) | 1 (1)
Hospitalized for shoulder surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hospitalized for attempted overdose (Psychiatric disorders) | 1 (1) | 1 (1)
Hospitalized for pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Emergency Department visit for chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Hospitalized for COVID-19 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Emergency Department visit for tremors and headache (Psychiatric disorders) | 0 (0) | 1 (1)
Emergency Department visit for high blood pressure (Cardiac disorders) | 1 (1) | 0 (0)
Hospitalized for broken hip (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hospitalized for knee replacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Project Life Force (N=101) | Treatment-As-Usual (N=106)
Emergency Department visit for back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Emergency Department visit for jaw pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Emergency Department visit for cough, headache, chills, fever (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Emergency Department visit for rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Increase in suicidal ideation/depression (Psychiatric disorders) | 1 (3) | 1 (1)
Challenges transferring inpatient programs (Social circumstances) | 1 (1) | 0 (0)
Loss of employment (Social circumstances) | 2 (2) | 1 (1)
Emergency Department visit for blood clot post surgical operation (Cardiac disorders) | 1 (1) | 0 (0)
Emergency Department visit for COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Emergency Department visit for substance withdrawl (Psychiatric disorders) | 0 (0) | 1 (1)
Emergency Department visit for leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Emergency Department visit for trouble breathing due to air quality (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Financial hardship and housing insecurity (Social circumstances) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Primarily, we experienced disruption in the planned procedures due to COVID-19 (e.g., necessitating a shift to remote treatment). This context limits the conclusions that can be drawn from this trial, as the in-person group setting was hypothesized to be an important mechanism of change and improvement in study outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2024-08-03): https://cdn.clinicaltrials.gov/large-docs/37/NCT03653637/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2025-05-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT03653637/SAP_001.pdf